CLINICAL TRIAL: NCT07205666
Title: The Eplontersen Pregnancy and Lactation Outcomes Study (EPPRO): A Descriptive Safety Study of Pregnant and Lactating Individuals and Their Offspring Exposed to Eplontersen
Brief Title: The Eplontersen Pregnancy and Lactation Outcomes Study
Acronym: EPPRO
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: D8451R00002
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Amyloidosis
Keywords: Eplontersen; pregnancy; Wainua; Wainzua
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of this DPSS is to describe the occurrence of pregnancy and maternal complications, adverse effects on the developing fetus and neonate, and adverse effects on the infant associated with exposure to eplontersen during pregnancy and/or lactation.

DETAILED DESCRIPTION:
Currently, there are no clinical studies of eplontersen use in pregnant individuals. Although it is expected that exposure to eplontersen during pregnancy or lactation is very rare, it is important to capture as many exposed cases as possible. This descriptive pregnancy safety study (DPSS) will add to the current body of knowledge regarding the safety of eplontersen exposure during pregnancy and lactation and maternal, fetal, and infant outcomes following exposure to eplontersen. The study is designed to fulfill health authorities' post-marketing requirements. This DPSS will analyze secondary data on cases of eplontersen-exposed pregnant and lactating individuals collected through a PRegnancy outcomes Intensive Monitoring (PRIM) enhanced pharmacovigilance (PV) approach utilizing AstraZeneca's PV Global Safety Database (PV-Argus). Data sources:

All eplontersen-exposed cases reported to AstraZeneca PV-Argus as notifiable events related to pregnancy and lactation; and cases reported from clinical trials, spontaneous post-marketing reports, post-marketing observational studies, patient-oriented programs, published literature, and personal communication by healthcare providers will be eligible for inclusion in the analysis. Data on eplontersen-exposed cases will be captured and processed using a pre-specified follow-up schedule and questionnaires. In case of missing data, there will be several attempts to collect data using all contact methods supplied by the reporters at the time of initial report.

Study size:

This DPSS is descriptive in nature, and a formal sample size calculation is not performed. Feasibility calculations indicate that the DPSS may capture five exposed pregnancies over the study period. Data analysis:

Analyses will be conducted in accordance with the study objectives, table/listing shells, and applicable guidelines. Demographics, medical and obstetric history, and disease characteristics will be summarized using descriptive statistics. The outcomes will be reported as a proportion and 95% confidence interval (if applicable) and calculated by dividing the number of cases of the outcome by the appropriate denominator for the particular outcome. If fewer than ten cases are reported, formal analyses will not be performed, and reporting will be limited to case narratives.

ELIGIBILITY:
Inclusion Criteria:

* all pregnancy and/or lactation cases with exposure to eplontersen and a diagnosis of an approved indication for treatment with eplontersen
* all adverse event reports in infants in the first 12 months of age that are or can be linked to pregnancy or lactation reports in individuals previously diagnosed with an approved indication and exposed to eplontersen during pregnancy or lactaction

Exclusion Criteria:

* all case reports considered invalid (i.e. minimum data is not provided at first report nor follow-up), or where reporter indicates that they do not wish to be contacted to obtain follow-up information, or the reporter/patient cannot be identified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant and/or lactating individuals
Study Population: The study population will include all PV reports of pregnant and/or lactating individuals diagnosed with an indication approved for use of eplontersen who administered at least one dose of eplontersen during pregnancy or lactation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2035-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
Major congenital malformations | November 2025 - December 2035
  All major congenital malformations diagnosed in utero, at birth or during the the first year of life. Considering the small number of patients anticipated to be included in this study, it is possible that only case narratives will be developed. However, if at least ten exposed pregnancies are reported, the data will be summarized quantitatively, using relevant measures. Major congenital malformation will be reported as numbers and proportions. When presented, the 95% confidence intervals (CIs) for proportion of the outcome of interest will be constructed using the exact (Clopper-Pearson) method.

SECONDARY OUTCOMES:
composite outcome of pregnancy and infant adverse outcomes ( except major congenital malformation | November 2025-December 2035
  pregnancy complications, spontaneous abortion, stillbirth, induced abortion, preterm birth, small for gestational age, postnatal growth deficiencies, infant development delay, neonatal mortality, infant mortality, as well as any other infant adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Myriam Alexander, PHD, Principal Investigator — AstraZeneca
Locations (1):
- Research Site, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The enhanced pharmacovigilance approach used in the study involves extraction of targeted safety questionnaire for pregnant or breastfeeding women exposed to eplontersen and reporting to AZ as part of routine pharmacovigilance

REFERENCES:
- [Result] Geissbuhler Y, Rezaallah B, Moore A. An alternative to product-specific pregnancy registries? PRIM; PRegnancy outcomes Intensive Monitoring. Reprod Toxicol. 2020 Jun;94:13-21. doi: 10.1016/j.reprotox.2020.03.004. Epub 2020 Mar 10. PMID 32169556